CLINICAL TRIAL: NCT03749408
Title: Effect of Addition of 0.5 Mol/L Mannitol to 0.5% Bupivacaine on IANB Success and Post-endodontic Pain in Mandibular Molars With Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Effect of Addition of Mannitol to Bupivacaine on IANB Success and Post-endodontic Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Safeya AbdelRahaman Hassan, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2012-12-24
Record Dates: First submitted 2018-11-15; First posted 2018-11-21 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Irreversible Pulpitis
Keywords: inferior alveolar nerve block; long-acting local anesthesia; bupivacaine; mannitol; symptomatic irreversible pulpitits
MeSH Terms: interventions — Bupivacaine; Mannitol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine plus mannitol (Active Comparator): 0.5% bupivacaine with 1:200,000 epinephrine plus 1.5 ml of 0.5 mol/L mannitol
  Interventions: Drug: bupivacaine plus mannitol
- bupivacaine alone (Experimental): 0.5% bupivacaine with 1:200,000epinephrine alone
  Interventions: Drug: bupivacaine alone

INTERVENTIONS:
Drug: bupivacaine plus mannitol — local anesthesia
  Other Names: vivacaine plus mannitol
  Arms: bupivacaine plus mannitol
Drug: bupivacaine alone — local anesthesia
  Other Names: vivacaine
  Arms: bupivacaine alone

SUMMARY:
Inferior alveolar nerve block using either 0.5% bupivacaine alone or in addittion to mannitol in patients with irreversible pulpitis in mandibular molars.

DETAILED DESCRIPTION:
Patients with irreversible pulpitis in mandibular molars will be selected according to the eligibility criteria and patients are then randomized to either using 0.5% bupivacaine alone or in addition to mannitol. Anesthetic success and postoperative pain will then be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients; age between 17-35 years old.
2. Males or Females.
3. Medically-free patients
4. Patients suffering from symptomatic irreversible pulpitis without apical periodontitis in mandibular molar teeth.
5. Positive patients' acceptance for participation in the study.

Exclusion Criteria:

* Patients who had any analgesic during proceeding 12 hours before the treatment.
* Teeth with necrotic, infected pulp, swelling or symptomatic apical periodontitis (apical abscess).
* Pregnant females.
* Patients with history of significant medical conditions (contraindication of mannitol use).
* Addiction
* Psycological disturbance.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity ranging from 0-10 where 0 means no pain, 10 the worst pain | 6 hours
  using pain scale ranging from 0-10 where 0 means no pain, 10 the worst pain
Postoperative pain intensity ranging from 0-10 where 0 means no pain, 10 the worst pain | 12 hours
  using pain scale ranging from 0-10 where 0 means no pain, 10 the worst pain
Postoperative pain intensity ranging from 0-10 where 0 means no pain, 10 the worst pain | 24 hours
  using pain scale ranging from 0-10 where 0 means no pain, 10 the worst pain
Postoperative pain intensity ranging from 0-10 where 0 means no pain, 10 the worst pain | 48 hours
  using pain scale ranging from 0-10 where 0 means no pain, 10 the worst pain
Postoperative pain intensity ranging from 0-10 where 0 means no pain, 10 the worst pain | 72 hours
  using pain scale ranging from 0-10 where 0 means no pain, 10 the worst pain

SECONDARY OUTCOMES:
Anesthetic success | 1 hour
  yes or no
lip numbness duration | 24 hours
  recorded in hours
Medication intake | 72 hours
  yes or no

IPD SHARING:
Plan to Share IPD: No